CLINICAL TRIAL: NCT02167737
Title: "ED-STEADI:" The Emergency Department Stopping Elderly Accidents, Deaths and Injuries Program (A Pilot Study)
Brief Title: The Emergency Department Stopping Elderly Accidents, Deaths and Injuries Program
Acronym: ED-STEADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Department of Emergency Medicine Research, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #PRO-00001450
Record Dates: First submitted 2014-06-14; First posted 2014-06-19 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Accidental Falls; Falling Injury; Other and Unspecified Fall on Same Level
Keywords: Accident Prevention; Accidental Falls; Geriatric Health Services; Gender Differences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bedside Decision Aid Group (Experimental): This arm will include study participants who are randomized to the group utilizing the bedside decision aid, which has hospital staff arrange fall-risk reduction interventions (e.g., home safety checks, exercise programs, vision checks, etc.).
  Interventions: Behavioral: Bedside Decision Aid
- Control Arm (Active Comparator): Participants in the control/comparator arm will experience the same study procedures with the exception of not using the Bedside Decision Aid and instead being given the Centers for Disease Control (CDC) brochure, "What You Can Do to Prevent Falls," and arranging for their own fall prevention strategies.
  Interventions: Behavioral: Control Arm

INTERVENTIONS:
Behavioral: Bedside Decision Aid — This group will have an initial FES and VES screening completed in the ED, the TUG test and Chair 30-Second Stand test, and the participant's risk of falling evaluated using our Bedside Decision worksheets. A study team member explains what subjects can do to decrease their risk of falling and discuss what mobility goals are the most important to them.
  Participants will receive a follow-up telephone call approximately six weeks after their discharge from the ED to collect self-reported data about goal completion, and then at four additional times--three, six, nine and 12 months--over the course of a year to collect self-reported data such as fall history.
  Arms: Bedside Decision Aid Group
Behavioral: Control Arm — This group will also have an initial FES and VES screening completed in the ED and the same two mobility tests (TUG and Chair 30-Second Stand). Study staff will advise subjects on how to take action to prevent falls and give them a brochure, "What YOU Can Do to Prevent Falls," from the CDC's "STEADI Tool Kit for Health Care Providers."
  Participants will receive a telephone call approximately six weeks after their discharge from the ED to collect self-reported data about goal completion, and then at four additional times--three, six, nine and 12 months--over the course of a year to collect self-reported data such as fall history.
  Arms: Control Arm

SUMMARY:
This study aims to determine if a bedside decision aid used in the ED for mechanical fall prevention can increase patient participation in management options that decrease their fall risk. Additionally, the investigators aim to determine if there are gender differences in patient choices in management options and accomplished goals inspired by the decision tool.

DETAILED DESCRIPTION:
This prospective, randomized controlled study will be conducted when there is a member of the research team available to consent patients at a Level I Trauma Center with approximately 90,000 annual ED visits across all age groups. Each potentially eligible patient will be identified by the research team and approached in the ED. Consented and enrolled patients will be assigned a study identification number and the enrollment documented by a member of the research team in the ED's electronic medical record after subjects are confirmed to meet inclusion and exclusion criteria. Subjects will be assigned randomly (by using a computer generated sequence) to either the control or intervention study arms.

Subjects in the control arm will have demographic data collected, a baseline Falls Efficacy Scale (FES) and Vulnerable Elders Survey (VES) screening completed and two STEADI Tool Kit mobility tests administered (the "TUG" [Timed Up and GO] and the 30-Second Chair Stand test). The FES and VES are validated surveys measuring fall concern and functional decline. The research team will advise them that they have a risk of falling as identified by inclusion criteria and that we are advising them to take action to prevent future falls. They will be given the brochure, "What YOU Can Do to Prevent Falls," that is standardized information recommended in the STEADI Tool Kit for Health Care Providers by the Centers for Disease Control (CDC).

Subjects in the active arm will also have demographic data collected, a baseline FES and VES screening completed, and two STEADI Tool Kit mobility tests administered (the "TUG" [Timed Up and GO] and the 30-Second Chair Stand test). Their risk of falling will be reviewed with them using a bedside decision aid indicating what they can do to decrease their risk. Particular attention will be given to personalizing their fall risk. The fall prevention management options will be presented in a value neutral fashion, along with the advantages and disadvantages of each option. They will have an opportunity to discuss what outcomes are the most important to them and choose the management options from the list provided that are the most valuable to them. Study and treatment team members will then work with this agreed upon selection to provide reliable intervention and outpatient follow up to improve the gains that can be realized in an integrated healthcare system. If the participant chooses to do their own home safety evaluation, they will be provided with a checklist to guide them in looking for hazards in their home and how to fix them. The patient will keep the original copy of their decision aid with their agreed-upon selected treatment options, and a copy of it will be placed in the subject's study file. All actions that are in response to the subject's selected plan (prescriptions, appointments, etc.) will also be documented in the study file.

Both groups will have phone follow-up at 6 weeks post ED visit, and then again at 3, 6, 9 and 12 months to collect self-reported data about goal completion and fall history. The last phone follow-up will include an exit FES and VES reassessment. All participants in both arms will have data collected about their inpatient and outpatient visits throughout the network during the study period to corroborate their self-report (e.g., occupational therapy, physical therapy visits, hospital admissions or ER visits for injuries related to a fall, etc.).

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* Be 65 years of age or older
* Be discharged home from the ED
* Be able to speak English.
* Be competent and able to give consent (not in critical condition, intoxicated or otherwise incapacitated)
* Have a mechanical fall risk as defined by one of the following:

Reports to have fallen in the last year Reports worrying about falling Admits they feel unsteady when standing or walking

Exclusion Criteria:

Patients must not:

* Be younger than 65 years old
* Be discharged from the ED to anywhere, but home (i.e., must not be discharged to family member's home, personal care facility, nursing home, group home, etc.)
* Be unable to speak English
* Be incompetent and unable to give consent (in critical condition, intoxicated or otherwise incapacitated)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of the bedside decision tool/worksheet | 12 months
  A single sheet bedside decision aid form/worksheet will be used to engage the patient in a discussion about fall prevention, the aim of which is to increase patient interest and participation in different management options that decrease fall risk. Patients will be followed up via phone calls re: their management option choices and how thorough/successful they were in completing them.

SECONDARY OUTCOMES:
Gender differences in use of the decision tool | 12 months
  Responses from the bedside decision tool choices will be grouped by gender to determine if men and women select different management options and/or have different patterns in completing them.

OTHER OUTCOMES:
Gender differences in fall management choices | 12 months
  Participants in *both* study arms will have phone follow-ups at the same time intervals to determine if men and women have different management option preferences and/or different patterns in completing them.

CONTACTS AND LOCATIONS:
Overall Officials: Marna R. Greenberg, DO, MPH, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Emergency Medicine Research, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD, just publish the study's results.